CLINICAL TRIAL: NCT03532178
Title: A Double-Blind, Randomized, Crossover Design Study To Compare The Rocuronium Reversal By Sugammadex To Succinylcholine For Electroconvulsive Therapy (ECT)
Brief Title: Comparison Of Rocuronium Reversal By Sugammadex To Succinylcholine For Electroconvulsive Therapy (ECT)
Acronym: CRoSSECT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: MISP#56343
Record Dates: First submitted 2018-04-03; First posted 2018-05-22 (Actual); Results first posted 2023-09-08 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-08

CONDITIONS: Neuromuscular Blockade
Keywords: Electroconvulsive Therapy, Neuromuscular Blockade
MeSH Terms: interventions — Sugammadex

STUDY DESIGN:
Intervention Model Description: The participants will be randomized to one of the two drug groups to start with, and will switch to the other group for the next treatment period. For the study, each participant will take two treatments in a random order: (1) rocuronium to be reversed by sugammadex, and (2) succinylcholine plus normal saline placebo.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The randomization of treatment groups will be blinded to the patients themselves, the psychiatrists and outcome assessors, except the anesthesiologists who will administer the drugs.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): rocuronium + sugammadex / succinylcholine + normal saline
  Interventions: Drug: Group A. "Muscle relaxant #1": rocuronium + sugammadex; "Muscle relaxant #2": succinylcholine +saline
- Group B (Experimental): succinylcholine + normal saline / rocuronium + sugammadex
  Interventions: Drug: Group B. "Muscle relaxant #2": succinylcholine +saline; "Muscle relaxant #1": rocuronium + sugammadex;

INTERVENTIONS:
Drug: Group A. "Muscle relaxant #1": rocuronium + sugammadex; "Muscle relaxant #2": succinylcholine +saline — The participants will be randomized to start with "Muscle relaxant #1" in the first study treatment, and will switch to "Muscle relaxant #2" in the second study treatment period.
  Other Names: Rocuronium: Zemuron. Sugammadex: Bridion. Succinylcholine: Suxamethonium
  Arms: Group A
Drug: Group B. "Muscle relaxant #2": succinylcholine +saline; "Muscle relaxant #1": rocuronium + sugammadex; — The participants will be randomized to start with "Muscle relaxant #2" in the first study treatment, and will switch to "Muscle relaxant #1" in the second study treatment period.
  Arms: Group B

SUMMARY:
The investigators propose to compare the recovery of neuromuscular blockade from rocuronium reversal by sugammadex to succinylcholine in ECT.

DETAILED DESCRIPTION:
The proposed study is a single center, randomized, double-blind (patients, psychiatrists and outcome assessor), cross-over clinical trial comparing the recovery of neuromuscular blockade from rocuronium with reversal of sugammadex to succinylcholine in participants receiving ECT. The primary outcome will be the measurement of time when the first train-of-four (TOF) twitch (T1) returns to 90% of baseline. The secondary aims are to document the safety (adverse event rates) of rocuronium/sugammadex compared to succinylcholine in ECT patients. The exploratory aims are to establish the perioperative efficacy and efficiency of sugammadex reversal of rocuronium in ECT procedures in comparison with succinylcholine.

ELIGIBILITY:
Inclusion Criteria:

* Eligible and scheduled for ECT
* Has the capacity to consent for the study

Exclusion Criteria:

* Any acute major organ failure in the last 30 days
* Any known or suspected neuromuscular disorders
* Any history of allergic reaction or intolerance to sugammadex, rocuronium, or succinylcholine
* Any conditions with severe renal impairment, including those requiring dialysis
* Anyone currently taking lithium
* Anyone currently taking hormonal contraceptives
* Anyone taking anti-coagulants, including vitamin K antagonists, unfractionated heparin, low molecular weight heparinoids, rivaroxaban, and dabigatran

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chanhung Lee, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Parnassus Campus, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lisanby SH. Electroconvulsive therapy for depression. N Engl J Med. 2007 Nov 8;357(19):1939-45. doi: 10.1056/NEJMct075234. No abstract available. PMID 17989386
- [Background] Fink M. What was learned: studies by the consortium for research in ECT (CORE) 1997-2011. Acta Psychiatr Scand. 2014 Jun;129(6):417-26. doi: 10.1111/acps.12251. Epub 2014 Feb 12. PMID 24571807
- [Background] Friedman S, Baker T, Gatti M, Simon G, Paskin S. Probable succinylcholine-induced rhabdomyolysis in a male athlete. Anesth Analg. 1995 Aug;81(2):422-3. doi: 10.1097/00000539-199508000-00040. No abstract available. PMID 7618742
- [Background] Iwatsuki N, Kuroda N, Amaha K, Iwatsuki K. Succinylcholine-induced hyperkalemia in patients with ruptured cerebral aneurysms. Anesthesiology. 1980 Jul;53(1):64-7. doi: 10.1097/00000542-198007000-00013. No abstract available. PMID 7386911
- [Background] Gijsenbergh F, Ramael S, Houwing N, van Iersel T. First human exposure of Org 25969, a novel agent to reverse the action of rocuronium bromide. Anesthesiology. 2005 Oct;103(4):695-703. doi: 10.1097/00000542-200510000-00007. PMID 16192761
- [Background] Ali HH, Utting JE, Nightingale DA, Gray C. Quantitative assessment of residual curarization in humans. Br J Anaesth. 1970 Sep;42(9):802-3. No abstract available. PMID 4248487
- [Background] Murphy GS, Brull SJ. Residual neuromuscular block: lessons unlearned. Part I: definitions, incidence, and adverse physiologic effects of residual neuromuscular block. Anesth Analg. 2010 Jul;111(1):120-8. doi: 10.1213/ANE.0b013e3181da832d. Epub 2010 May 4. PMID 20442260
- [Background] Lee C, Jahr JS, Candiotti KA, Warriner B, Zornow MH, Naguib M. Reversal of profound neuromuscular block by sugammadex administered three minutes after rocuronium: a comparison with spontaneous recovery from succinylcholine. Anesthesiology. 2009 May;110(5):1020-5. doi: 10.1097/ALN.0b013e31819dabb0. PMID 19387176
- [Background] Mirzakhani H, Guchelaar HJ, Welch CA, Cusin C, Doran ME, MacDonald TO, Bittner EA, Eikermann M, Nozari A. Minimum Effective Doses of Succinylcholine and Rocuronium During Electroconvulsive Therapy: A Prospective, Randomized, Crossover Trial. Anesth Analg. 2016 Sep;123(3):587-96. doi: 10.1213/ANE.0000000000001218. PMID 26967896
- [Background] Sparr HJ, Vermeyen KM, Beaufort AM, Rietbergen H, Proost JH, Saldien V, Velik-Salchner C, Wierda JM. Early reversal of profound rocuronium-induced neuromuscular blockade by sugammadex in a randomized multicenter study: efficacy, safety, and pharmacokinetics. Anesthesiology. 2007 May;106(5):935-43. doi: 10.1097/01.anes.0000265152.78943.74. PMID 17457124
- [Background] Kadoi Y, Hoshi H, Nishida A, Saito S. Comparison of recovery times from rocuronium-induced muscle relaxation after reversal with three different doses of sugammadex and succinylcholine during electroconvulsive therapy. J Anesth. 2011 Dec;25(6):855-9. doi: 10.1007/s00540-011-1236-y. Epub 2011 Sep 24. PMID 21947754

RESULTS

PARTICIPANT FLOW:
Period: First Period
Arm/Group | Group A | Group B
Started | 23 | 21
Completed | 22 | 17
Not Completed | 1 | 4
Not completed — Withdrawal by Subject | 1 | 3
Not completed — technical issues in data collection Technical issues | 0 | 1
Period: Second Period
Arm/Group | Group A | Group B
Started | 22 | 17
Completed | 21 | 15
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Technical issues | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 23 | 21 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 19 | 37
  >=65 years | 5 | 2 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 22
  Male | 13 | 9 | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 2 | 2
  Hispanic or Latino | 3 | 0 | 3
  Africa American | 0 | 0 | 0
  American Native | 0 | 0 | 0
  unreported | 0 | 1 | 1
  More than 1 race | 0 | 0 | 0
  White | 20 | 18 | 38

OUTCOME MEASURES:

1. Primary Outcome: Recovery Time of T1 to 90% Baseline
Description: The time of neuromuscular recovery from sugammadex 4mg/kg dose reversal rocuronium at 0.6 mg/kg compared with traditionally used succinylcholine in electroconvulsive therapy (ECT).
Time Frame: 30 minutes
Population: Subjects completed the two periods with each study medication
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Muscle Relaxant #1: rocuronium 0.6 mg/kg + reversal with sugammadex 4 mg/kg
- Muscle Relaxant #2: succinylcholine 1.0 mg/kg + reversal with normal saline as the placebo agent
Arm/Group | Muscle Relaxant #1 | Muscle Relaxant #2
Number analyzed (Participants) | 36 | 36
minutes | 6.79 (2.08) | 10.97 (3.06)

2. Secondary Outcome: Number of Participants With Treatment or Emergent Adverse Events of the Drugs
Description: To document the side-effect profiles of sugammadex reversal of rocuronium and succhinylcholine in the ECT patient population
Time Frame: 24 hours after the procedure
Measure: Count of Participants; unit: Participants
Groups:
- Rocuronium + Sugammadex: rocuronium 0.6 mg/kg + reversal with sugammadex 4 mg/kg
- Succinylcholine + Normal Saline: succinylcholine 1.0 mg/kg + reversal with normal saline as the placebo agent
Arm/Group | Rocuronium + Sugammadex | Succinylcholine + Normal Saline
Number analyzed (Participants) | 40 | 40
Participants
  Nausea | 1 | 3
  Myalgia | 1 | 2
  Headache | 7 | 9

ADVERSE EVENTS:
Time Frame: 24 hours following the treatment
Arm/Group | Rocuronium + Sugammadex | Succinylcholine + Normal Saline
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 9/40 | 14/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rocuronium + Sugammadex (N=40) | Succinylcholine + Normal Saline (N=40)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Headache (Nervous system disorders) | 7 (7) | 9 (9)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) — muscle soreness
Pain and swelling at i.v. catheter site (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-11-03): https://cdn.clinicaltrials.gov/large-docs/78/NCT03532178/Prot_SAP_000.pdf
  • Informed Consent Form (2020-12-10): https://cdn.clinicaltrials.gov/large-docs/78/NCT03532178/ICF_001.pdf